CLINICAL TRIAL: NCT05832658
Title: Efficacy of Game-Based EMG-Biofeedback Therapy in Post-Stroke Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Bulent Alyanak, Research assistant, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-68869993-000-1019202
Record Dates: First submitted 2023-04-16; First posted 2023-04-27 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Stroke; Dysphagia; Surface Electromyography; Biofeedback; Swallowing Disorder
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMG-Biofeedback (Experimental): Mendelsohn maneuver and effortful swallow exercise will be applied through game-based emg-biofeedback to patients with post-stroke dysphagia.
  Interventions: Device: With EMG-Biofeedback; Behavioral: Usual Care
- Classic Therapy (Active Comparator): Mendelsohn maneuver and effortful swallow exercise with only verbal feedback will be applied to patients with post-stroke dysphagia.
  Interventions: Behavioral: Without EMG-Biofeedback; Behavioral: Usual Care

INTERVENTIONS:
Device: With EMG-Biofeedback — Once a day for a total of 15 sessions, the Mendelsohn maneuver will be performed for 15 minutes and the effortful swallow maneuver will be performed for 15 minutes with game-based emg-biofeedback.
  Arms: EMG-Biofeedback
Behavioral: Without EMG-Biofeedback — Once a day for a total of 15 sessions, the Mendelsohn maneuver will be performed for 15 minutes and the effortful swallow maneuver will be performed for 15 minutes with only verbal feedback.
  Arms: Classic Therapy
Behavioral: Usual Care — Patient and family education will be provided by the investigator. In addition, each patient will be evaluated and oral motor exercises and thermal tactile stimulation will be given to each patient when necessary.

SUMMARY:
This study aims to determine the effectiveness of game-based biofeedback application via surface electromyography in patients with post-stroke dysphagia. The same treatment interventions will be applied with and without biofeedback, and thus the contribution of adding biofeedback to the treatment will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. History of hemorrhagic or ischemic stroke longer than 3 months
2. Being over the age of eighteen
3. Level ≤ 6 on the Functional Oral Intake Scale (FOIS)
4. Post-stroke onset of swallowing complaints
5. Ability to communicate with the patient and carry out the given commands
6. Mini mental test evaluation ≥ 24 points
7. Absence of concomitant serious systemic disease (unregulated hypertension, decompensated heart failure, malignancy, infection, pacemaker, epilepsy, etc.)
8. Detection of pathology in the oropharyngeal phase of swallowing in videofluoroscopic evaluation
9. Not taking any swallowing-related treatment in the last 3 months

Exclusion Criteria:

1. History of neoplastic disease and/or radiotherapy to the head and neck region
2. Having additional musculoskeletal disease or non-stroke neurologic disease that may cause swallowing disorders
3. Unable to communicate or carry out commands
4. Inability to maintain head-holding balance
5. Patients with severe pathology in bolus formation or delivery of the bolus to the pharynx during the oral swallowing phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-05-07 (Actual); Primary Completion 2023-10-14 (Actual); Study Completion 2023-10-14 (Actual)

PRIMARY OUTCOMES:
Gugging Swallowing Screen (GUSS) | From baseline to the end of the treatment ( 3 week)
  It is used to determine the severity of dysphagia and the risk of aspiration in patients with acute stroke. It is evaluated out of 20 points. It recommends videofluoroscopy as an advanced examination for patients with a score of less than 20.
Functional Oral Intake Scale (FOIS) | From baseline to the end of the treatment ( 3 week)
  7 point scale from 1-7. Higher number indicated increased amount and normality of oral intake.
Penetration Aspiration Scale (PAS) | From baseline to the end of the treatment ( 3 week)
  Videofluoroscopic evaluation is performed. It is an 8-point scale. The higher the number, the greater the increase in penetration/aspiration. 1 means no penetration and no aspiration. 8 means there is aspiration and there is no patient response.
Functional Dysphagia Scale (FDS) | From baseline to the end of the treatment ( 3 week)
  Videofluoroscopic evaluation is performed. It is a total of 100 points scale. A higher score indicates more severe dysphagia.
Dysphagia Outcome and Severity Scale (DOSS) | From baseline to the end of the treatment ( 3 week)
  Videofluoroscopic evaluation is performed. It is a 7-point scale. A score of 6 and 7 represents normal swallowing, a score of 5 represents mild dysphagia, a score of 2 to 4 represents moderate dysphagia, and a score of 1 represents severe dysphagia.
Dysphagia Handicap Index (DHI) | From baseline to the end of the treatment ( 3 week)
  Dysphagia Handicap Index (DHI) is a self-assessment questionnaire which consists of 25 statements to examine three aspects of dysphagia patients' quality of life (QoL): functional, physical, and emotional. The patient can get a maximum score of 100 points.A higher score indicates a more severe swallowing disorder.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No